CLINICAL TRIAL: NCT02655042
Title: A Long-term Follow-up Study to Evaluate the Safety and Efficacy of RCT-01 in Men and Women With Unilateral, Chronic Achilles Tendinosis
Brief Title: Long-Term Follow-up of the Safety and Efficacy of RCT-01 in Men and Women With Unilateral, Chronic Achilles Tendinosis
Acronym: ReaCT-X
Status: Withdrawn | Type: Observational
Why Stopped: Study conduct does not meet corporate objectives of sponsor
Sponsor: RepliCel Life Sciences, Inc. (Industry)
Collaborators: Syreon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: RCT-01-002-2015
Record Dates: First submitted 2016-01-05; First posted 2016-01-13 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Tendinosis; Tendinopathy
MeSH Terms: conditions — Tendinopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- RCT-01: Participants in previous clinical trial that received blinded injection of RCT-01
- Placebo: Participants in previous clinical trial that received blinded injection of placebo

SUMMARY:
The primary purpose of this study is to assess the long-term safety profile of RCT-01 injections as compared to placebo injections. This study will also measure the long-term impact these injections will have on tendon structure and function and the symptoms of Achilles tendinosis.

This is study is designed to follow participants who have completed participation in a clinical trial where they received injections of either RCT-01 or placebo in the Achilles tendon. No clinical interventions will be performed as part of study procedures.

The day of study entry (Visit 1) will be coordinated with the participant's final visit in the earlier clinical trial. All participants will return to the clinic for repeat assessments of their Achilles tendinosis and overall health 6, 12 and 18 months after study entry. Furthermore, they will complete 'telephone visits'; during which they will report information on their overall health; 3, 9, and 15 months after study entry. Total duration of patient participation is approximately 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Participation in a clinical trial designed to evaluate RCT-01 treatment for chronic Achilles tendinosis. Participants must complete the final study visit in the earlier trial prior to participation in this clinical trial.
* Willingness to provide written informed consent for participation in the study, attend all study visits and complete all procedures required by this protocol.

Exclusion Criteria:

* The presence of any condition that, in the investigator's opinion would impact participant safety and/or a participant's ability to complete all study related procedures. (e.g., psychiatric illness, drug addiction, alcoholism, etc.)

NOTE: age limits not specifically set in this trial as entry into current trial based on qualification/completion of previous clinical trial where age rage of participants was explicitly stated.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have completed participation in a clinical trial to evaluate the safety and efficacy of injections of RCT-01.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 24 months post-injection
  Comparison of the safety profile between RCT-01/placebo treatment groups. The safety profile is defined by the incidence, relationship to treatment, severity and seriousness of adverse events.

SECONDARY OUTCOMES:
Victorian Institute of Sport Assessment - Achilles (VISA-A) questionnaire | 24 months post-injection
  pain on palpation and pain on loading (running/jumping)
Modified Tegner Activity Scale | 24 months post-injection
SF-36 questionnaire | 24 months post-injection
  quality of life questionnaire
Tendon condition (appearance) | 24 months post-injection
  Ultrasound imaging will be utilized to measure region and relative location (from calcaneus) of damage and overall tendon size (in mm)
Tendon condition (blood flow) | 24 months post-injection
  Ultrasound imaging will be utilized to measure blood flow (vascularization) within the tendon. Defined on ordinal scale
Tendon condition (fibrillar pattern) | 24 months post-injection
  Fibrillar pattern observed during ultrasound imaging of tendon structure will be graded on ordinal scale.
Tendon condition (presence of abnormalities) | 24 months post-injection
  Presence/absence of intratentinous calcification, observable tears, and irregularities in calcaneus bone structure will be noted during ultrasound imaging.

CONTACTS AND LOCATIONS:
Overall Officials: D R Lloyd-Smith, MDCM, Principal Investigator — University of British Columbia
Locations (1):
- Alan McGavin Sports Medicine Centre, Vancouver, British Columbia, Canada

REFERENCES:
- See also: RepliCel Corporate Website — http://www.replicel.com